CLINICAL TRIAL: NCT02956551
Title: Neoantigen-primed DC Vaccine Therapy for Refractory Non-small Cell Lung Cancer
Brief Title: Personalized DC Vaccine for Lung Cancer
Acronym: SKLB1608
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sichuan University (Other)
Responsible Party: Principal Investigator, Zhen-Yu Ding, Professor, Sichuan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SKLB1608
Record Dates: First submitted 2016-11-01; First posted 2016-11-07 (Estimated); Last update posted 2018-05-31 (Actual); Status verified 2018-05

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: advanced non-small cell lung cancer; cell based therapy; safety; clinical efficacy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — lentiviral minigene vaccine of COVID-19 coronavirus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- cell_therapy (Experimental): tumor neoantigen primed DC vaccines are administrated, 2-week interval, totally 5 times
  Interventions: Biological: DC vaccine

INTERVENTIONS:
Biological: DC vaccine — subcutaneous administration

SUMMARY:
The study is aimed to the test the efficacy and safety of neoantigen-primed dendritic cell (DC) cell vaccine therapy for refractory non-small cell lung cancer.

DETAILED DESCRIPTION:
Patients with pathological confirmed non-small cell lung cancer with no standard treatment are enrolled. The patients fails in previous at least 2 lines of chemotherapy and 1 line of targeted therapy where applicable. This is a prospective exploratory trial. Patients' rebiopsy tumor tissues are subsequent to whole exosome sequencing and possible neoantigens are identified. DC is in vitro primed with synthesized peptides. Both adverse events and responses are recorded.

ELIGIBILITY:
Inclusion Criteria:

* pathologically confirmed non-small cell lung cancer
* failed in previous standard chemotherapy and targeted therapy
* anticipated life time > 3month
* Karnofsky performance status 0-1
* rehabilitate from previous therapy
* adequate organ functions

Exclusion Criteria:

* mixed histological types
* tumor emergency
* abnormal coagulation condition
* contagious diseases, such as hepatitis B virus, hepatitis C virus, human immunodefficiency virus, tuberculosis infection
* concomitant tumors
* immunological co-morbidities

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-11-30 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-06-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 3 months after the last administration of cells
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0

SECONDARY OUTCOMES:
objective response rate | through study completion, an average of 1 year
  Number of participants with objective responses as assayed by RECIST 1.1

CONTACTS AND LOCATIONS:
Overall Officials: Zhen-Yu Ding, Prof, Principal Investigator — Sichuan University
Locations (1):
- China West Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided